CLINICAL TRIAL: NCT03758911
Title: Perspectives on the Adolescent, Young Adult, and Adult Experience as Donors for Their Parent Undergoing Haploidentical Bone Marrow Transplants
Brief Title: Perspectives on Bone Marrow Donors Who Donate for Their Parent
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: J16127; IRB00111131 (Other: JHM IRB); 2016-03p (Other: Palliative Care Research Consortium)
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Bone Marrow Transplant
Keywords: bone marrow; stem cell; donor; interview

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bone marrow/blood stem cell donors: Participants underwent a one time semi-structured telephone interview to understand the perspectives of bone marrow/stem cell donors experience, including how family dynamics impacted participants' decision to donate and identifying unique supportive care needs of bone marrow/stem cell donors.
  Interventions: Other: Semi-structured Interview

INTERVENTIONS:
Other: Semi-structured Interview

SUMMARY:
The purpose of this pilot study is to explore the role of family function on decision-making for bone marrow donors who donated for their parent, and to assess the unique supportive care needs of these participants. Semi-structured interviews were conducted with participants to identify overarching themes of the donation experience.

ELIGIBILITY:
Inclusion Criteria:

* Donated bone marrow or peripheral blood stem cells for their parent in the past 1-6 months
* Willing to participate in mandatory audio recorded telephone interview
* Able to participate in interview without assistance
* Must be English speaking
* Transplant recipient (parent) must be living

Exclusion Criteria:

* Unable to provide oral consent for participation (for minors- unable to obtain parental consent and/or oral assent from child for participation)

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants included adolescents, young adults, or adults who had donated bone marrow or peripheral blood stem cells for their parent in the past 1 - 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Themes influencing donors' decision-making as assessed by words used during interview responses | Day 1
  Words/terms are extracted from interviewer responses and associated to key themes that influence participant's decision-making process. A codebook is used to reference these words/terms

CONTACTS AND LOCATIONS:
Overall Officials: Nina D Wagner-Johnston, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Undecided